CLINICAL TRIAL: NCT06274593
Title: Study of OCT Peripapillary Angiography in Patients With Advanced Glaucoma
Acronym: OGA
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AP_JBD_MJ_003
Record Dates: First submitted 2024-02-14; First posted 2024-02-23 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Glaucoma
Keywords: glaucoma; OCTa; OCTrnfl
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: OCT — Peripapillary angiography (OCT) at baseline and each year during 3 year

SUMMARY:
Glaucoma is a chronic disease of the optic nerve, characterized by progressive loss of nerve cells in the retina, leading to progressive loss of peripheral and central vision. There are in fact several types of glaucoma, which is the world's second leading cause of blindness after cataracts, and the leading cause of irreversible blindness.

To date, to our knowledge, there is no work analyzing the progression of angiographic OCT in patients with glaucoma.

The main aim of this study is to compare the 3-year progression rate of 3 examinations in advanced glaucoma patients: one functional (visual field) and two anatomical (OCTa and OCTrnfl).

DETAILED DESCRIPTION:
Glaucoma is a chronic disease of the optic nerve characterized by progressive loss of nerve cells in the retina, leading to progressive loss of peripheral and central vision. There are in fact several types of glaucoma, which is the world's second-leading cause of blindness after cataracts and the leading cause of irreversible blindness.

The pathophysiology and loss of retinal ganglion cells are partly explained by 2 main theories:

* biomechanical theory, which takes into account the forces and deformations of the optic nerve linked to IOP (intraocular pressure) and to the anatomy of the optic nerve head, particularly at the level of the cribriform plate (a zone of deformable weakness surrounded by a rigid scleral shell),
* the vascular theory, explained by abnormalities in the vascularization of the optic nerve and retina.

Optical coherence tomography angiography (OCTa) is a relatively new imaging method that has been on the market for around ten years.

It is a non-invasive method that provides qualitative and quantitative information on retinal vascularization and the optic nerve head. The movement of red blood cells is used as a contrast medium to differentiate blood vessels from static tissue.

In glaucoma, changes in the peripapillary vascular plexus (around the optic nerve head) can be observed and are topographically correlated with visual field and peripapillary nerve fiber deficits.

One of the challenges in monitoring glaucoma patients lies in detecting the progression of the disease with the help of various complementary examinations, including the visual field, peripapillary nerve fiber OCT (RNFL), and more recently, OCTa.

The visual field is used to detect areas of vision deficit (peripheral or sometimes central), known as scotomas, and to monitor their evolution. RNFL OCT measures the thickness of the optic nerve (in micrometers) in its various quadrants. OCTa measures vascular density, also by quadrant, around the optic nerve head.

A deterioration in any of these parameters can help guide therapeutic management by modifying medical treatment or proposing surgery to lower intraocular pressure in the affected eye.

One of the difficulties in monitoring glaucoma patients lies in detecting optic nerve thinning in patients with advanced optic nerve damage. It is now well known that at an advanced stage of the disease, measurement of optic nerve thickness on RNFL OCT can reach a "floor" effect: residual non-neuronal tissue limits the usefulness of detecting changes in neuronal tissue, and disease progression can only be detected by visual field monitoring.

Vascular density measured on OCTa appears to reach a plateau effect in a delayed manner compared with measurements obtained on peripapillary OCT (RNFL) and could enable better monitoring of disease progression in patients with advanced glaucoma.

Indeed, a new objective follow-up criterion measured with OCTa in clinical practice for patients with uninterpretable OCTrnfl would be a valuable tool for assessing the rate of glaucoma progression in these patients and thus defining the rate of monitoring and the decision to intensify treatment in the event of progression. This is all the more important as the treatments available for glaucoma are sometimes invasive (drainage devices, surgery, etc.). Assessing the benefit-risk balance therefore requires objective data for these patients.

To date, to our knowledge, there are no studies analyzing the evolution of OCT angiography in glaucoma patients.

The main aim of this study is to compare the 3-year progression rate of 3 examinations in advanced glaucoma patients: one functional (visual field) and two anatomical (OCTa and OCTrnfl).

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 and over
* Patient with glaucoma followed in the ophthalmology department of Nantes University Hospital
* mean visual field deficit (MD) >10dB

Exclusion Criteria:

* Retinal vascular pathology (moderate to severe non-proliferative diabetic retinopathy, complicated diabetic retinopathy, OVCR/OBVR, OACR/OBAR, NOIAA...) Non-glaucomatous optic neuropathy, neurological pathology leading to visual field deficit (stroke with HLH, quadranopsia, chiasmatic Sd...)
* PPR (retinal PanPhotocoagulation), retinal cerclage
* Retinal pathology leading to visual field impairment (e.g. retinitis pigmentosa)
* AMD and other macular pathologies that can lead to central visual field deficits
* Significant environmental disorders impairing retinal imaging (e.g. active uveitis, dense cataract)
* Loss of fixation point preventing visual field formation Pregnant or breast-feeding women
* Protected adults under guardianship or curatorship
* with unreliable visual fields (false positives and false negatives > 33%)
* with an uninterpretable OCTrnfl or OCTa (artifact, low quality score)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients followed at Nantes University Hospital for advanced glaucoma (MD>10dB in visual field) who had peripapillary angiography OCT, OCTrnfl and visual field at their follow-up consultation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-04-27 (Actual); Primary Completion 2027-04-27 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Compare the progression of vascular density (VD) in advanced glaucoma patients. | 3 year
  Progression of peripapillary vascular density (VD) (in percent) per sector (8 sectors) with 3-year follow-up.
Compare the progression of peripapillary retinal nerve fiber (RNFL) thickness) in advanced glaucoma patients. | 3 year
  Progression of peripapillary nerve fiber thickness (RNFL, in µm) per sector (8 sectors) with 3-year follow-up.
Compare the progression of visual field in advanced glaucoma patients. | 3 year
  Progression of visual field deficit (in dB) by sector (8 sectors) with 3-year follow-up

SECONDARY OUTCOMES:
CV-OCTrnfl correlation study and CV-OCTa correlation study on measurements made at inclusion and on measurements made during follow-up | 3 years
  Study of the correlation between CV-OCTrnfl and correlation between CV-OCTa (mean in µm)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Nantes, Nantes
  - Jean-Baptiste Ducloyer, Nantes

IPD SHARING:
Plan to Share IPD: No